CLINICAL TRIAL: NCT05752084
Title: Jaundice Predisposes to the Incidence of Nosocomial Infection in Egyptian Patients With Cirrhosis: A Cohort Study
Brief Title: Bilirubin Increases the Risk of Nosocomial Infection in Cirrhotic Patients
Acronym: {bilirubin}
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Khadija Ahmed Mhrose Glal, assistant lecturer, Tanta University
Other Study IDs: TantaUu
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Nosocomial Infection
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: the group that develops Nis during the study
- group 2: the group doesn't develop NIs

SUMMARY:
Nosocomial infection (NIs) is a major challenge in healthcare facilities and has been associated with prolonged hospital stay as well as increased morbidity and mortality.

This research aimed to estimate the impact of acute decompensation (AD) consequences on the successive risk of nosocomial infections (NIs) and the go after outcome.

DETAILED DESCRIPTION:
Cirrhosis is the 14th most widespread cause of mortality worldwide [1], cirrhosis can take one of the following forms: compensated and decompensated phases [2]. The latter is related to subsequent complications such as ascites, hepatic encephalopathy (HE), gastrointestinal hemorrhage (GIH), jaundice, or spontaneous bacterial peritonitis (SBP) [2]. Decompensated cirrhosis is a common cause of frequent hospital admission and high fatality rate [3]. Patients with cirrhosis and decompensation have bacterial translocations (BT) and immune deterioration [4]. Therefore, they are susceptible to getting infections and septic shock [5]. On the other hand, the infection can worsen the course of cirrhosis and hasten the progression of related morbidities with a subsequent increase in death rate owing to its ability to accelerate organ failure [6]. For cirrhotic patients, the occurrence of NIs is an essential standpoint [7]. Several studies on cirrhotic patients revealed that the incidence of NIs is much higher in patients with cirrhosis and thus worsens the prognosis [8,9]. Recent studies showed that around 30 to 50% of bacterial infections (BIs) in patients with decompensated cirrhosis are NIs which is related to a higher risk of acute-chronic liver failure (ACLF), severe sepsis, and mortality [10-12].

Nevertheless, current studies have not clarified how decompensation differentially predisposes to the occurrence of NIs and affects the outcomes. Henceforth, this study aimed to assess the incidence of NIs in cirrhosis with differential decompensation consequences, the bond between the type of decompensation at admission and the progress of NIs, and the synergism between decompensation and subsequent NIs on the outcome.

ELIGIBILITY:
Inclusion Criteria:

* cirrhotic patients both sex

Exclusion Criteria:

* pregnancy
* lactation
* HCC

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients were diagnosed with cirrhosis based on liver biopsy. Decompensation was defined as acute deterioration in liver function accompanied with acute onset of complications such as ascites, HE, GIH, BIs, or jaundice at the time of hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
occurrence of nosocomial infection | 1 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No